CLINICAL TRIAL: NCT00937833
Title: Randomized Controlled Trial Examining the Return of Urinary Continence After Robot-assisted Radical Prostatectomy With or Without a Urethrovesical Sling
Brief Title: Return of Continence Following Robot-Assisted Radical Prostatectomy With or Without a Urethrovesical Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-015; 350017
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Incontinence; Prostate Cancer
Keywords: prostate cancer; prostatectomy; incontinence
MeSH Terms: conditions — Urinary Incontinence; Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Urethrovesical Sling (Experimental): Surgisis Male Sling placed at the time of prostatectomy
  Interventions: Procedure: Prostatectomy; Device: Surgisis Male Sling
- Control (Active Comparator): Prostatectomy
  Interventions: Procedure: Prostatectomy

INTERVENTIONS:
Procedure: Prostatectomy
Device: Surgisis Male Sling
  Arms: Urethrovesical Sling

SUMMARY:
The purpose of this study is to determine the impact of an absorbable urethrovesical sling on the post-operative return of urinary continence after robot-assisted radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have organ confined prostate cancer.
* Patients must have PSA< 15.
* Patients must have clinical stage prostate cancer < cT3.
* Patients must be scheduled for robot assisted transperitoneal laparoscopic radical prostatectomy.
* Patients must be able to provide written informed consent and HIPAA authorization for release of personal health information.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Patients must not have previously undergone transurethral resection, laser therapy, microwave therapy, radiofrequency ablation, or other surgery of the prostate.
* Patients must not have previously undergone incision of urethral stricture or incision of bladder neck contracture.
* Patients must not have previously been diagnosed with urethral stricture, bladder neck contracture or urinary incontinence.
* Patients must not have previously been diagnosed with atonic bladder or neurogenic bladder.
* Patients must not have significant pre-operative voiding symptoms as defined by an American Urologic Association symptom score of greater than 19.
* Patients must not have a prior history of radiation to the pelvis.
* Patients must not have persistent bacteriuria that cannot be cleared, as demonstrated by a negative urinalysis or urine culture, within 1 month of surgery.
* Patients must not have allergies to pig tissue or pig products or have religious or cultural objection to the use of pig tissue.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandru Sundaram, MD, Principal Investigator — Indiana Cancer Pavilion
Locations (2):
- United States (2):
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Urology of San Antonio Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Urethrovesical Sling: Surgisis Male Sling: The SurgiSIS Biodesign, a urethrovescial sling, is placed at the time of prostatectomy.
- Control: No sling placed at the time of prostatectomy
Period: Overall Study
Arm/Group | Urethrovesical Sling | Control
Started | 73 | 77
Completed | 58 | 60
Not Completed | 15 | 17
Not completed — Protocol Violation | 1 | 2
Not completed — Procedure delayed; enrollment closed | 0 | 1
Not completed — Lost to Follow-up | 10 | 8
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Population: 147 patients were treated with the study procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Urethrovesical Sling | Control | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (6.1) | 60.6 (7.1) | 60.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 73 | 74 | 147

OUTCOME MEASURES:

1. Primary Outcome: Number of Continent Patients Post Prostatectomy
Time Frame: 1 Month
Measure: Number; unit: participants
Arm/Group | Urethrovesical Sling | Control
Number analyzed (Participants) | 67 | 68
participants | 37 | 32

ADVERSE EVENTS:
Arm/Group | Urethrovesical Sling | Control
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/74
Other Adverse Events (participants affected / at risk) | 0/73 | 0/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urethrovesical Sling (N=73) | Control (N=74)
Hospitalization (Renal and urinary disorders) | 2 (2) | 0 (0)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0)
Intervention to prevent impairment (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days